A Retrospective Study To Evaluate The Safety And Efficacy Of A Neucleoside-Sparing Regimen Of Darunavir, Ritonavir AND Dolutegravir

NCT03198884

8/2/2019

A Retrospective Study To Evaluate The Safety and Efficacy Of A Neucleoside-Sparing Regimen Of Darunavir, Ritonavir And Dolutegravir

John Verna, PA-C, AAHIVS | SIHF Healthcare, Sauget, IL

Stephen Austin, MS | Washington University in St. Louis, St. Louis, MO

### Background

Aging with HIV infection is a relatively new phenomenon and investigators are only beginning to understand its implications for clinical care and for our understanding of aging more generally. Several sequelae of aging with HIV have been identified, including increased cardiovascular risk, bone loss, and renal dysfunction. Various antiretrovirals have been implicated in contributing to or exacerbating these conditions, most specifically the nucleoside reverse transcriptase inhibitors (NRTI) class. Despite the approval of various new pharmaceutical compounds over the last few years, the NRTI class remains limited in safe therapeutic options. The most commonly used NRTI, tenofovir, has been implicated in numerous studies causing and/or contributing to renal disorders in persons with HIV [1,2,3]. In addition, data from the D:A:D study has shown in increased risk of cardiovascular disease (CVD) among patients receiving treatment for HIV and that certain medications appear to be associated with that risk, including the NRTI abacavir [4]. HIV therapy is life-long and providers have opted to use nucleosidesparing regimens to minimize these toxic effects. The purpose of this study is to determine the realworld efficacy and safety of a nucleoside-sparing regimen of darunavir 800 mg, ritonavir 100 mg, and dolutegravir 50 mg by mouth once daily. While not well studied, this two-drug regimen was chosen for its lack of drug-drug interactions [5], predictable pharmacokinetic profile [6] and exceptional tolerability [7,8,9].

### Methods

We conducted a retrospective chart review of approximately 400 HIV+ patients receiving treatment at SIHF Healthcare, an urban diverse FQHC to identify those who were receiving a NRTI-sparing regimen of DRV and DTG. Subjects were included if they were ≥ 18 years of age, receiving DRV/r QD + DTG QD for ≥ 24 weeks, and had laboratory data through 48 weeks of follow up. Subjects were excluded if they received a regimen of darunavir/ritonavir in combination with dolutegravir for <24 weeks duration, if they received darunavir/ritonavir + DTG + NRTI's, missed more than five doses over two weeks prior to study visit or if there was missing laboratory data for ≥2 or more study time points. The primary endpoints evaluated were the percent of patients with an RNA <50 copies/mL at 48 weeks after initiation of the once daily two-drug regimen, as well as, the change in serum creatinine from baseline to 48 weeks. Main secondary endpoints included changes from baseline in CD4+ cell counts, incidence and severity of adverse events and, analysis of RNA and serum creatinine at time points 24, 36 and 48 weeks.

The percent of patients with an RNA <50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure. Change in mean serum creatinine from baseline was analyzed using Wilcoxon signed rank test.

Change in mean CD4+ cell counts from baseline was analyzed using a paired t-test. All analyses used a p-value of less than or equal to 0.05 as significant. Statistical analyses were performed using R software, version 3.4.3.

### Results

The Mean age of the cohort was 51 yrs and had an average of 12.5 years of HIV seropositivity. Table 1. The cohort had a mean baseline CD4+ of 485 with an RNA of 20K copies. Table 2. Of note, 55% of study subjects had a viral load of > 50 copies at baseline. 95% of study subjects at week 48 met the primary endpoint of < 50 copies/mL (P-value 0.002), 95%CI [2.24, NA]. Figure 1. The lone failure was due to missing data. Also, there were no significant differences in serum creatinine from baseline to 48 weeks (p = 0.5753). Figure 2. However, at week 24, one study subject did not have data (serum creatinine) in window. There were no significant changes in CD4+ cell count from baseline at time points 24, 36 or 48 weeks. Figure 3.

Table 1

| Descr | Descriptive Stats - Demographics | | | | |
|---|---|---|---|---|---|
| | N | % | | | |
| Gender | | | A | Age in years | |
| Female | 8 | 40% | | Mean (SE) | 51.05 (0.96) |
| Male | 12 | 60% | | Median | 53.00 |
| Race | | | | Range | 37.00 - 61.00 |
| Black | 15 | 75% | | std | 8.20 |
| White | 5 | 25% | H | IIV in years | |
| | | | | Mean (SE) | 12.54 (0.98) |
| | | | | Median | 9.50 |
| | | | | Range | 0.25 - 32.00 |
| | | | | std | 8.79 |
| | | | | Veight in Pounds | |
| | | | | Mean (SE) | 160.30 (4.04) |
| | | | | Median | 157.00 |
| | | | | Range | 106.00 - 244.0 |
| | | | | std | 33.77 |

Table 2

| escriptive Stats – CD4 and Viral Loa | | | | |
|---|---|---|---|---|
| Complive States CD4 and viral Loa | | | | |
| Viral Load | Baseline | Week 24 | Week 36 | Week 48 |
| N | 20 | 19 | 14 | 19 |
| Missing=Failure | 0 | 1 | 6 | 1 |
| Mean (SE) | 20458 (12389.4) | 10232 (9559.583) | 33.57 (12.82) | 22.63 (1.50) |
| Median | 95.0 | 20 | 20.00 | 20.00 |
| Range | 20.0 - 207720.0 | 20 -1820101 | 20.00 - 200 | 20.00 - 40.00 |
| SD | 55407.07 | 41669.26 | 47.98 | 6.53 |
| CD4 Count | Baseline | Week 24 | Week 36 | Week 48 |
| N | 20 | 20 | 14 | 20 |
| Missing=Failure | 0 | 0 | 6 | 0 |
| Mean (SE) | 485.1 (67.0) | 453.9 (67.22) | 428.1 (67.95) | 455.7 (64.98) |
| Median | 458.5 | 379.5 | 376.0 | 428.5 |
| Range | 24.0 – 1011.0 | 93.0 – 1145.0 | 112.0 – 877.0 | 70.0 – 1142.0 |
| SD | 299.41 | 300.64 | 254.24 | 290.56 |

Figure 1



Figure 2



Figure 3



### **Adverse Events**

As per the study protocol, an adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product.

Of note, there was no treatment-emergent resistance detected or virological failures in any of the subjects. Common side effects reported by patients were insomnia (30%), diarrhea (20%) and headache (15%). There were no adverse events that led to discontinuation of the study regimen. Table 3.

Table 3 [10]

| Patient ID | Adverse | Severity | Relationship to Study | Action Taken | Suspected study |
|---|---|---|---|---|---|
| | Event | | Product | | drug: DRV/r or DTG |
| #2 | Diarrhea | Grade 1 | Possible | None | DRV/r |
| #4 | Insomnia | Grade 1 | Possible | None | DTG |
| #6 | Insomnia | Grade 1 | Possible | None | DTG |
| #7 | Headache, | Grade 1 | Possible | None | Both |
| | Diarrhea | | | | |
| #8 | Headache, | Grade 1 | Possible | None | Both |
| | Diarrhea | | | | |
| #9 | Insomnia | Grade 1 | Possible | None | DTG |
| #10 | Insomnia | Grade 1 | Possible | None | DTG |
| #14 | Insomnia | Grade 1 | Possible | None | DTG |
| #15 | Insomnia | Grade 1 | Possible | None | DTG |
| #20 | Headache, | Grade 1 | Possible | None | Both |
| | Diarrhea | | | | |

## Adverse Drug Reaction

As per study protocol, an adverse drug reaction (ADR) is defined as a response to a medicinal product that is noxious and unintended.

Of note, no adverse drug reactions were reported during this study.

# Serious Adverse Event

As per study protocol, this is defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product or is otherwise medically important.

Of note, no serious adverse events were reported during this study.

Finally, no female subject (40% or 8/20 subjects) became pregnant during the 48 weeks of the study.

#### Discussion

The results show that after 48 week of darunavir 800 mg, ritonavir 100 mg and dolutegravir 50mg by mouth once daily, patients were able to maintain virologic suppression and there were no discontinuations due to adverse events.

Clinically, this regimen may be beneficial for patients who experience side effects with other antiretroviral therapy or for those who struggle with adherence issues as this is a once daily regimen. However, there are several limitations to this research. Due to the small sample size and data selection from a single center, it is difficult to extrapolate the results to the general HIV population. Additionally, using snapshot analysis to evaluate efficacy can be flawed as it may not reflect the true response characteristics over the whole treatment phase.

Toxicities associated with antiretroviral compounds are drug-class specific. A commonly used NtRTI was tenofovir disoproxil fumarate (TDF). This compound is known to affect renal function and bone mineral density (BMD). In 2016, the Food And Drug Administration (FDA) approved a TDF pro-drug, tenofovir alafenamide [11]. Switching to this compound was associated with statistically significant efficacy and safety advantages over TDF [12].

The NEAT study (NEAT001/ANRS143) found that the regimen of raltegravir in combination with darunavir/ritonavir was about equal to a triple drug regimen of tenofovir/emtricitabine in combination with darunavir/ritonavir in terms of efficacy and safety in treatment naïve patients [13]. However, subjects with CD4 counts below 200 cells/µL and viral loads above 100,000 copies/mL did not do as well

A second study was SWORD-1/SWORD-2 which evaluated the N(t)RTI sparing, dual-drug regimen of once-daily dolutegravir plus rilpivirine vs. current antiretroviral regimen (CAR). The authors found that at week 48, the regimen of dolutegravir plus rilpivirine was non-inferior to CAR and showed a safety profile consistent with its components, supporting the use of this two-drug regimen to maintain HIV suppression [14].

### Conclusion

In this study the combination of darunavir/ritonavir in combination with dolutegravir yielded high rates of virologic suppression. While some patients experienced adverse events known to be associated with darunavir or dolutegravir, all adverse events were low grade and did not require discontinuation of treatment or alteration in dose

### References

- 1. Morlat P, Vivot A, Dauchy F, et al. Antiretroviral drugs and incidence of chronic kidney disease, ANRS CO3 Aquitaine cohort (2004-2008). Program and abstracts of the 6th IAS Conference on HIV Pathogenesis, Treatment and Prevention: July 17-20, 2011; Rome, Italy. Abstract WEPBD0104
- 2. Goicoechea M, Liu S, Best B, et al. Greater tenofovir-associated renal function decline with protease inhibitor-based versus nonnucleoside reverse-transcriptase inhibitor-based therapy. J Infect Dis. 2008; 197: 102-108
- 3. Gallant JE, Moore RD. Renal function with the use of a tenofovir-containing initial antiretroviral regimen. AIDS. 2009; 23:1971-1975
- 4. Friis-Møller N, Sabin CA, Beber R, et al. Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med. 2003 Nover 20; 349(21): 1993-2003. Erratum in: N Engl J Med. 2004 Feb 26; 350(9): 955.
- 5. Lexicomp Online, Lexicomp® Drug Interactions, Hudson, Ohio: Wolters Kluwer Clinical Drug Information, Inc.; 2018
- 6. Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV. Department of Health and Human Services USA, Washington, DC; 2018
- 7. Prezista® [package insert]. Titusville, NJ: Janssen Therapeutics, Division of Janssen Products, LP; 2006
- 8. Norvir® [package insert]. North Chicago, IL: AbbVie Inc.; 1996
- 9. Tivicay® [package insert]. Research Triangle Park, NC: ViiV Healthcare; 2013
- 10. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 July 2017
- 11. Descovy® [package insert]. Foster City, CA: Gilead Sciences, Inc; 9/2017
- 12. DeJesus E, Haas B, Segal-Maurer, etal. Superior Efficacy and Improved Renal and Bone Safety After Switching from a Tenofovir Disoproxil Fumarate-to a Tenofovir Alafenamide-Based Regimen Through 96 Weeks of Treatment. AIDS Research and Human Retroviruses. 2018 Apr;34(4):337-342
- 13. Raffi F, Babiker AG, Richert L, et al. Ritonavir-boosted darunavir combined with raltegravir or tenofovir-emtricitabine in antiretroviral-naïve adults infected with HIV-1: 96 week results from the NEAT001/ANRS143 randomized non-inferiority trial. Lancet. 2014 Nove 29;384(9958):1942-51.
- 14. Llibre JM, Hung CC, Castelli F, et al. Efficacy, safety, and tolerability of dolutegravir-rilpivirine for the maintenance of virological suppression in adults with HIV-1: phase 3, randomized, non-inferiority SWORD-1 and Sword-2 studies. Lancet. 2018 Mar 3;391(10123):839-849.